CLINICAL TRIAL: NCT01292109
Title: Compliance and Efficacy in the Use of PICOPREP for Bowel Cleansing
Brief Title: A Study of PICOPREP in Patients Needed to Clean the Bowel Prior to X-ray Examination, Endoscopy or Surgery.
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999169 CS03
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Bowel Cleanliness
Keywords: endoscopy; colonoscopy; preparation for surgery
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICOPREP®
  Interventions: Drug: sodium picosulphate

INTERVENTIONS:
Drug: sodium picosulphate — Sodium picosulphate (PICOPREP®) taken by participant prior to X-ray examination, endoscopy or surgery.
  Other Names: PICOPREP®

SUMMARY:
The study serves as a confirmation of safety, tolerance and efficacy of PICOPREP in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving PICOPREP® for bowel evacuation prior to endoscopy or surgery

Exclusion Criteria:

* Patients in which prescription of PICOPREP® is contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients about to undergo X-ray examination, endoscopy or surgery.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Documentation of use PICOPREP in everyday practice | Day 0 - 2

SECONDARY OUTCOMES:
Participant satisfaction and compliance after bowel cleansing | Days 0-2
Participants with adverse events reported by frequency and severity | Days 1-2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (3):
- Czechia (3):
  - University Hospital, Ostrava - Poruba
  - University Hospital, Pilsen
  - Iscare - Prague 7, Prague